# Are There Patterns and Trends in Patient Engagement When Participating in Renal Cell Carcinoma Clinical Trials?

This is an Informed Consent Form For Renal Cell Carcinoma Patients in <a href="Power Clinical Trial's">Power Clinical Trial's</a> Observational Study

Date: October 15, 2023

Grasping the Significance of This Informed Consent Document

Engaging with this paperwork suggests your potential qualification for involvement in an exclusive observational clinical investigation tailored to patients with renal cell carcinoma. This comprehensive manual outlines the fundamental aims of the study, the detailed execution plan, and the diverse ramifications, covering both beneficial and potentially negative outcomes. Before making any decisions, thoroughly understanding the specifics of your potential participation is vital, and seeking advice from a trusted source can provide crucial perspectives. If any part of this material appears perplexing or if you have any questions, rest assured that the researcher is available to offer clarifications.

Recognizing the Importance of Clinical Trials for Renal Cell Carcinoma

Renal cell carcinoma is a type of kidney cancer that originates in the lining of the proximal convoluted tubule, a part of the small tubes in the kidney that filter waste from the blood and produce urine. It is the most common type of kidney cancer in adults and accounts for approximately 90% of cases.

Clinical trials with a special focus on renal cell carcinoma are essential in evaluating the safety and effectiveness of new therapies for this condition. These trials serve as crucial

mechanisms to determine whether new drugs excel beyond traditional treatments, providing substantial evidence to endorse their broader use.

What makes this study unique is its primary concentration on the personal experiences of individuals facing renal cell carcinoma, actively participating in a clinical trial that involves medicinal interventions. The main objective is to meticulously analyze trial completion rates and voluntary withdrawals among this specific cohort of patients.

#### Immersing Yourself in Observational Clinical Trials

Engagement in this medical trial involves immersion in an observational study, an essential facet of clinical research meticulously crafted to gather insights through discreet monitoring of patients while upholding their treatment plans.

Researchers will solely observe your journey, meticulously evaluating the outcomes of your condition without implementing any alterations. This trial design is instrumental in enhancing our comprehension of the intrinsic progression of a specific medical ailment and its implications for those afflicted by it. Your active involvement in this observational study plays a pivotal role in advancing the boundaries of medical knowledge and driving improvements in the care provided to individuals grappling with the same issue.

Understanding the Distinctiveness of This Study from Other Renal Cell Carcinoma Clinical Trials

Recognizing the unique features of this research investigation is imperative. It functions solely on an observational basis, indicating that your involvement will not include any specific therapies or interventions. To make an informed decision about potential participation in a clinical trial, it is crucial to comprehend the array of renal cell carcinoma clinical research, encompassing interventional studies where participants undergo diverse treatment regimens.

Arriving at an informed decision about your potential participation in a clinical trial requires an active approach involving research and comparison of different trials. Resources like Clinicaltrials.gov and similar platforms offer abundant information about renal cell carcinoma research. Furthermore, Power's specialized online platform provides a comprehensive catalog of ongoing renal cell carcinoma clinical trials actively seeking volunteers. Empowered with thorough research and a comprehensive

understanding of various clinical trial categories, you can confidently determine your participation.

## Ensuring the Confidentiality of Your Information

As this research project unfolds, ensuring the complete confidentiality of your data remains of paramount importance. It is imperative to avoid including any personal or identifiable information in your questionnaire responses to maintain your anonymity. The research team is dedicated to fortifying the protection of your privacy. However, it's important to acknowledge that certain legal circumstances might arise, compelling the disclosure of personal data.

## Your Voice in Clinical Trial Surveys: An Invitation to Participate

We extend a warm invitation to actively share your insights as part of this observational clinical study. Engaging in this endeavor involves the periodic completion of surveys, each requiring approximately 20-30 minutes of your time. Additionally, we have structured quarterly check-in calls to ensure a comprehensive understanding throughout your involvement in the trial.

It's crucial to emphasize that your participation in the survey phase of the trial is entirely voluntary. You retain the autonomy to answer select questions or complete the entire questionnaire. Moreover, should you choose, you possess the liberty to withdraw from the trial at any point. Recognizing the personal nature of enrolling in a clinical trial, our commitment lies in providing the necessary support, respecting your privacy, and aiding in your decision-making process throughout the trial.

## Envisioned Gains and Impact

While immediate benefits may not be immediately discernible for participants in this observational clinical research, their involvement holds the potential to leave a significant mark on the medical community. The information derived from participants will be instrumental in refining future strategies for reaching out to individuals with renal cell carcinoma, potentially broadening the scope of medical investigation. Those who embark on this journey have the power to ignite substantial changes in medical research, potentially shaping the landscape for future renal cell carcinoma patients.

## **Understanding Potential Health Risks**

While clinical trials have made remarkable advancements, it is crucial to understand the potential health risks that participants may face, particularly in studies evaluating novel medications.

Nonetheless, our observational clinical research takes a distinctive approach, minimizing these risks by refraining from the use of experimental drugs in participants. Rather, our primary focus is on vigilant monitoring and evaluation of outcomes, aiming to prevent any unnecessary health hazards.

## **Encouraging Diversity in Clinical Studies**

A multitude of online platforms are ready to facilitate your active involvement if you are motivated by an insatiable curiosity to delve into the intricate domain of diversity within clinical trials.

Whether your goal is to grasp the complexities of the challenges and potentials linked to clinical trial diversity or to broaden your personal insights, the following resources can serve as valuable tools:

Motazedian, Pouya, Thais Coutinho, and F. Daniel Ramirez. "Female representation in clinical studies informing atrial fibrillation guidelines: have we built a house of cards?." Canadian Journal of Cardiology 38, no. 6 (2022): 709-711.

Bird, Chloe E. "Women's representation as subjects in clinical studies: a pilot study of research published in JAMA in 1990 and 1992." Women and health research: Ethical and legal issues of including women in clinical studies 2 (1994): 151-173.

## Acknowledgment of Informed Consent

I hereby acknowledge that I have devoted sufficient time to understanding and internalizing the contents of the informed consent form. This understanding has been attained through either self-examination or with the assistance of a trusted individual

who has expounded its key points to me. All of my concerns and queries have been fully addressed to my complete satisfaction.

I am fully cognizant that my participation in this study is entirely voluntary, and I retain the exclusive right to retract my consent without being obliged to offer justifications or assume any financial liabilities. It has been made clear to me that a duplicate of this informed consent form will be provided for my personal records.

After thorough consideration and careful review of all the materials provided to me, I hereby provide my consent to participate in this study, signifying my informed and self-reliant decision.

| Participant Name |
|-----------------------|
| Participant Signature |
| Date |

Verification by Informed Consent Facilitator

I verify that I engaged in a comprehensive conversation with the participant, meticulously unraveling the intricacies encompassed in this written material. My objective was to ensure that the participant fully grasped the primary study objectives, employed methodologies, potential risks and benefits, and other critical components of the renal cell carcinoma clinical trial.

The participant was provided ample opportunity to raise questions, express concerns, and seek clarification. It is crucial to underscore that the participant's involvement in this study is entirely voluntary, and they retain the unimpeded right to withdraw at any time, for any reason, without incurring any financial obligations.

| Subsequent to the participant's agreement, a carefully preserved duplicate of this written document was provided, serving as a repository for their specific information. |
|---|
| Printed Name of Assisting Researcher |
| Signature of Assisting Researcher |
| Date |